CLINICAL TRIAL: NCT04970940
Title: An Open-label, Multiple Dose, Crossover Study to Evaluate the Drug-drug Interaction Between AJU-A51R1 and AJU-A51R2 in Healthy Volunteers
Brief Title: The Drug-drug Interaction Study of AJU-A51R1 and AJU-A51R2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20DM10201
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence 1 (Experimental): * Period 1: Treatment A(AJU-A51R1: Farxiga 1 Tab., Q.D., single dose, for 5 days)
  * Wash-out for 7 days
  * Period 2: Treatment B(AJU-A51R2: Trajenta 1 Tab., Q.D., single dose, for 11 days)
  * Period 3: Treatment C(AJU-A51R1 1 Tab. and AJU-A51R2 1 Tab., Q.D., co-administration for 5 days)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — AJU-A51R1: Farxiga 1 Tab., Q.D., single dose, for 5 days
  Other Names: Period 1
Drug: Treatment B — AJU-A51R2: Trajenta 1 Tab., Q.D., single dose, for 11 days
  Other Names: Period 2
Drug: Treatment C — AJU-A51R1 1 Tab. and AJU-A51R2 1 Tab., Q.D., co-administration for 5 days
  Other Names: Period 3

SUMMARY:
To evaluate a pharmacokinetic drug interaction between AJU-A51R1 and AJU-A51R2 in healthy male volunteers.

DETAILED DESCRIPTION:
This study is to investigate drug-drug interaction between AJU-A51R1 and AJU-A51R2.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals whose age is over 19 and under 65 years old when visiting for initial screening test.
2. Body mass index(BMI) between 17.5~30.5 kg/m^2 and the body weight must be over 55 kg(men) or 45 kg(women) (Body mass index (BMI) = weight (kg) / height (m)^2) .
3. Individuals with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area.
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening after examined through hematology test and blood chemistry analysis, urinary test, the electrocardiogram (ECG), and etc.
5. The participants must be volunteered and sign in an informed consent document proven by Chonbuk National University IRB before joining a study to show that he was given informed the purpose of tests and the special characteristics of drugs.
6. Individuals who agreed proper contraception during the study
7. The participants must have an ability and willingness to participate throughout the entire trials.

Exclusion Criteria:

1. Individuals with a medical evidence or a history (excluding dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune disease.
2. Individual who had a history of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy).
3. Individual who had following results after examination(a. ALT or AST > twice higher than Upper limit of normal value).
4. Individual Who constantly intake 210 g/week of alcohol within 6 months of the screening. (a cup of beer (5%) (250 mL) = 10 g, a shot of soju (20%) (50mL) = 8 g, a glass of wine (12%) (125 mL) = 12g).
5. Individual whose blood pressure < 90 or ≥160(systolic blood pressure) or < 50 or ≥ 100(diastolic blood pressure).
6. Individuals who had been administered investigational product(s) from other clinical study or bioequivalence study within 180 days prior to the first dose of this study(except when subject have not taken investigational product(s)).
7. Individual who had a medical history of alcohol and drug abuses.
8. Individual who had taken a drug that has a control of metabolic rate (activation or inhibition) in 30 days before the first taking of clinical testing drug.
9. Individual who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders.
10. A person who is not determined unsuitable to participate in this test by the researchers.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
AUCτ of AJU-A51R1 and AJU-A51R2 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Area Under Curve tau
Css,max of AJU-A51R1 and AJU-A51R2 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Cmax, steady state

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, Principal Investigator — Jeonbuk University Hospital
Locations (1):
- Min-gul Kim, Jeonju, Korea, South Korea